CLINICAL TRIAL: NCT00259818
Title: An Open-Label Phase I Dose Escalation Study of Intravenous Infusion of Tetra-O-Methyl Nordihydroguaiaretic Acid (EM-1421) in Subjects With Refractory Malignant Tumors
Brief Title: Dose Escalation Study of EM-1421 for the Treatment of Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erimos Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-1421 #101
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Cancer
Keywords: Refractory; Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — terameprocol

INTERVENTIONS:
Drug: EM-1421

SUMMARY:
This is a Phase I, dose escalation study of EM-1421 administered by intravenous infusion (IV) for five consecutive days every 28 days to patients with solid tumors refractory to current therapies. There have been no previous human studies of intravenous (into one's vein) EM-1421 treatment; however, lab research (research in test tubes and/or animals) suggests that EM-1421 has shown some activity against tumors in animals. This activity in animal models suggests that EM-1421 may be a useful chemotherapy for human cancer.

The primary objective of this study is to determine the safety and maximum tolerated dose of EM-1421 given by intravenous infusion. The efficacy of the treatment will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age.
* Subjects with documented evidence of cancer with clinically evaluable disease. Cancer can be recurrent after primary treatment with surgery, radiation therapy, and/or chemotherapy and may include those patients for whom no standard or curative therapy exists.
* Measurable tumor by imaging (computed tomography [CT] per Response Evaluation Criteria in Solid Tumors [RECIST] criteria).
* Life expectancy of at least 3 months in the Investigator's opinion.
* Negative pregnancy test, if in women of childbearing potential, within one week of starting therapy.
* Subjects who have provided written informed consent to participate in the study.
* ECOG performance status of 0, 1, or 2.
* Absolute neutrophil ≥ 1500 cells/µL, hemoglobin ≥ 9 gm/dl, platelets ≥ 100,000/µL, ALT/AST ≤ 3 x ULN (upper limit of the normal range) unless involved with tumor then < 5 x ULN, bilirubin ≤ 1.5 x ULN, and creatinine ≤ 1.5 x ULN.

Exclusion Criteria:

* Women who are pregnant or breast-feeding (women of child-bearing potential must have a negative serum pregnancy test within one week of entering the study.)
* Women of child-bearing potential who are unwilling to use two medically acceptable forms of contraception during the course of the study (surgical sterilization, approved hormonal contraceptives, or barrier method with spermicide).
* Treatment with a prior investigational agent within 28 days of entering the study.
* Subjects unable to comply with the study requirements.
* Subjects with a known sensitivity to any of the study medication components.
* Prior chemotherapy, radiation therapy, or surgery for the primary tumor within 28 days of dosing and/or has not recovered from prior therapy toxicities - with the exception of non-experimental chronic hormone therapy for currently progressive metastatic prostate cancer. However, local radiation to a site of symptomatic disease will be acceptable if it has been completed at least 14 days prior to study drug initiation and subjects have recovered from all treatment-related side effects.
* Subjects exhibiting any of the following: a marked baseline prolongation of QT/QTc interval (repeated demonstration of a calculated QTc interval > 450), a history of additional risk factors for torsades de pointes (TdP) (e.g., heart failure, hypokalemia, family history of long QT syndrome), and subjects unable or unwilling to refrain from using medications that are known to prolong the QT/QTc ratio during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-12; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Safety
Maximum tolerated dose

SECONDARY OUTCOMES:
Pharmacokinetic parameters
Pharmacodynamic parameters
Anti-tumor activity of regimen
Feasibility of regimen

CONTACTS AND LOCATIONS:
Overall Officials: Neil Frazer, MB — Erimos Pharmaceuticals
Locations (3):
- United States (3):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Albert Einstein College of Medicine, The Bronx, New York
  - Sarah Cannon Cancer Center, Nashville, Tennessee